CLINICAL TRIAL: NCT03725410
Title: Clinical Evaluation of the Safety and Performance of Using Multi-Polar RF and PEMF Technologies for the Treatment of Symptoms Associated With Vulvovaginal Atrophy
Brief Title: Multi-polar RF and PEMF for Treatment of Symptoms Associated With Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CS1017
Record Dates: First submitted 2018-10-26; First posted 2018-10-31 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-02

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venus Fiore Study Treatment (Active Comparator): Study treatment consists of delivering radiofrequency (RF) and pulsed electromagnetic fields (PEMF) internally to the vagina (50 - 70% for up to 15 minutes), externally to the labia (10 - 35% for up to 10 minutes) and externally to the mons pubis (10 - 35% for up to 15 minutes).
  Interventions: Device: Venus Fiore Study Treatment
- Venus Fiore Sham Treatment (Placebo Comparator): Sham treatment consists of delivering radiofrequency (RF) and pulsed electromagnetic fields (PEMF) internally to the vagina (1% for up to 15 minutes), externally to the labia (1% for up to 10 minutes) and externally to the mons pubis (1% for up to 15 minutes).
  Interventions: Device: Venus Fiore Sham Treatment

INTERVENTIONS:
Device: Venus Fiore Study Treatment — Study treatment consists of delivering radiofrequency (RF) and pulsed electromagnetic fields (PEMF) internally to the vagina (50 - 70% for up to 15 minutes), externally to the labia (10 - 35% for up to 10 minutes) and externally to the mons pubis (10 - 35% for up to 15 minutes).
  Arms: Venus Fiore Study Treatment
Device: Venus Fiore Sham Treatment — Sham treatment consists of delivering radiofrequency (RF) and pulsed electromagnetic fields (PEMF) internally to the vagina (1% for up to 15 minutes), externally to the labia (1% for up to 10 minutes) and externally to the mons pubis (1% for up to 15 minutes).
  Arms: Venus Fiore Sham Treatment

SUMMARY:
This is a multicenter, single-blind, randomized, sham-controlled study utilizing the Venus Fiore™ (MP)2, a table-top device designed to deliver multi-polar RF energy and pulsed electromagnetic fields for use in dermatological and general surgical procedures to temporarily improve blood circulation and to induce modification of collagen structure, neocollagenesis and angiogenesis for the treatment of symptoms associated with vulvovaginal atrophy.

DETAILED DESCRIPTION:
Multicenter, single-blind, randomized, sham-controlled study of multi-polar radio-frequency (RF) and pulsed electro-magnetic field (PEMF) technologies for the treatment of symptoms associated with vulvovaginal atrophy. The study will enroll up to 106 subjects requesting treatment of symptoms of vulvovaginal atrophy (vaginal dryness, decreased lubrication during sexual activity, decreased elasticity, irritation, discomfort during intercourse and discomfort of the vaginal and vulvar tissues in general) in order to have 88 subjects complete the study. Subjects will be randomized in a 1:1 ratio to either multi-polar RF and PEMF technologies or sham treatment and will receive a total of three internal and external treatments with the Venus Fiore™ (MP)2 device at four-week intervals. Study treatment will be administered as per the parameter recommendations as set out in the Venus Fiore™ (MP)2 user manual. Subjects will be followed up at three and six months after their initial treatment. Analysis will be performed on all subjects who receive at least one treatment. Three- and six-month outcomes from the active arm will be compared to data from the sham arm.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female subjects, ≥ 19 years of age, requesting treatment of vulvovaginal tissue for improvement of symptoms associated with vulvovaginal atrophy
2. Baseline FSFI score <27.
3. At least one full-term vaginal delivery (of more than 36 weeks gestation) completed at least one year before study enrollment.
4. Able to read, understand and voluntarily provide written Informed Consent.
5. Able and willing to comply with the treatment/follow-up schedule and requirements.
6. Sexually active in a monogamous relationship.
7. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study, and have a negative Urine Pregnancy test at baseline.
8. Negative Papanicolaou (Pap) Smear Cytology Test within 3 months prior to enrollment.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the course of study.
2. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Having a permanent implant in the treated area (e.g. intrauterine device).
4. Prior use of collagen, fat injections and/or other methods of skin augmentation (enhancement with injected or implanted material) in the treated area within 4-6 weeks of the initial treatment or during the course of the study.
5. Use of retinoids such as oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study.
6. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
7. Open laceration, abrasion or bleeding of any sort on the area to be treated.
8. Active sexual transmitted disease (STD) (e.g. genital Herpes Simplex, condylomata) or vaginosis.
9. Chronic vulvar pain or vulvar dystrophy.
10. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications, including corticosteroids, 6 months prior to and during the course of the study.
11. Having any form of active cancer at the time of enrollment and during the course of the study.
12. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the treatment, or healing process.
13. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria.
14. Mentally incompetent or evidence of active substance or alcohol abuse.
15. Having any stage 3-4 cystocele, rectocele, enterocele paravaginal defect or major pelvic organ prolapse beyond the hymenal ring.
16. Unstable dosages of medications such as antihypertensives or psychotropics that are known to affect sexuality.
17. Skin piercing in the treatment area.
18. Tattoos in the treatment area.
19. Prior skin treatment with laser in the treated area within 6 months of the initial treatment or during the course of treatment.
20. Prior ablative resurfacing procedure in the treated area with laser or other devices within 12 months of the initial treatment or during the course of treatment.
21. History of keloid formation or poor wound healing in a previously-injured skin area.
22. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only human females have labia, a mons pubis and a vagina.
Enrollment: 81 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Vaginal Health Index (VHI) | Three months after initial treatment
  Proportion of subjects in the active arm as compared to the proportion of the subjects in the sham arm assessed as having improvement in the Vaginal Health Index (VHI) score.
Vaginal Health Index (VHI) | Six months after initial treatment
  Proportion of subjects in the active arm as compared to the proportion of the subjects in the sham arm assessed as having improvement in the Vaginal Health Index (VHI) score.
Vaginal Mucus | Three months after initial treatment
  Report the microscopic changes in vaginal mucus in the study treatment group as compared to the sham treatment group.
Vaginal Mucus | Six months after initial treatment
  Report the microscopic changes in vaginal mucus in the study treatment group as compared to the sham treatment group.
Vaginal pH | Three months after initial treatment
  Report the microscopic changes in vaginal pH in the study treatment group as compared to the sham treatment group.
Vaginal pH | Six months after initial treatment
  Report the microscopic changes in vaginal pH in the study treatment group as compared to the sham treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, PhD, Study Director — Venus Concept Ltd.
Locations (2):
- IRCCS Policlinico S. Matteo, Pavia, Italy
- Institute Palacios, Madrid, Spain